CLINICAL TRIAL: NCT04199598
Title: An Open-label, Single-center, Randomized, 4-period, Single Dose, Crossover Study to Assess the Relative Bioavailability of Abediterol Inhaled Via Two Different Nebulizers and Via Dry Powder Inhaler in Healthy Subjects.
Brief Title: Relative Bioavailability Study With Abediterol Administered Via Three Different Inhalation Devices in Healthy Volunteers.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate has been taken by the Sponsor. The decision is not due to safety concerns but reflects business prioritizations of the company.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D6541C00001
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Open-label; Long-acting beta-2 agonist; COPD; Bioavailability; Phase 1; Abediterol; Healthy subjects; Crossover
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 5-(2-((6-(2,2-difluoro-2-phenylethoxy)hexyl)amino)-1-hydroxyethyl)-8-hydroxyquinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment A (test product): Abediterol (2.4 μg) (Experimental): Randomized subjects will receive single dose treatment of Abediterol nebuliser solution for inhalation via PARI LC SPRINT nebulizer following an overnight fast of at least 8 hours
  Interventions: Drug: Abediterol (2.4 μg)
- Treatment B (Test Product): Abediterol (4.8 μg) (Experimental): Randomized subjects will receive single dose treatment of Abediterol nebuliser solution for inhalation via PARI LC SPRINT nebulizer following an overnight fast of at least 8 hours
  Interventions: Drug: Abediterol (4.8 μg)
- Treatment C(Test Product):Abediterol(2.4 μg) (Experimental): Randomized subjects will receive single dose treatment of Abediterol nebuliser solution for inhalation via OMRON NE-C900-E nebulizer following an overnight fast of at least 8 hours
  Interventions: Drug: Abediterol (2.4 μg)
- Treatment D (Reference Product): Abediterol (2.5 μg) (Experimental): Randomized subjects will receive single dose treatment of Abediterol (as napadisylate) inhalation powder via dry powder inhaler (DPI) following an overnight fast of at least 8 hours
  Interventions: Drug: Abediterol (2.5 μg)

INTERVENTIONS:
Drug: Abediterol (2.4 μg) — 2.4 μg (delivered dose) abediterol via PARI LC SPRINT nebuliser
  Arms: Treatment A (test product): Abediterol (2.4 μg)
Drug: Abediterol (4.8 μg) — 4.8 μg (delivered dose) abediterol via PARI LC SPRINT nebuliser
  Arms: Treatment B (Test Product): Abediterol (4.8 μg)
Drug: Abediterol (2.4 μg) — 2.4 μg (delivered dose) abediterol via OMRON NE-C900-E nebuliser
  Arms: Treatment C(Test Product):Abediterol(2.4 μg)
Drug: Abediterol (2.5 μg) — 2.5 μg (nominal dose) abediterol via DPI, reference
  Arms: Treatment D (Reference Product): Abediterol (2.5 μg)

SUMMARY:
The study is intended to assess the relative bioavailability of 2 different abediterol nebulised formulations (test) and the dry powder formulation (reference). The study results will provide information on the pharmacokinetic (PK) profile following use of the 3 devices to be used in further clinical development.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, 4-period, single-dose, single-center, crossover study with a William's design in healthy subjects (males).

The study will comprise:

1. A screening period of maximum 28 days;
2. Four treatment periods during which subjects will be resident prior to the evening meal the night before dosing with abediterol (Day -1) until at least 48 hours following dosing for collection of PK samples; discharged on the morning of Day 3; and
3. A final safety post-treatment visit within 14 days after the last administration of abediterol.

There will be a minimum washout period of 14 days between each treatment period.

Each subject will be involved in the study for approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures.
2. Healthy male subjects aged 18 - 45 years, inclusive, with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 18 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
4. Subject is able to understand and communicate in German.
5. Willing and able to comply with all required study procedures.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other conditions (e.g., including Gilbert's syndrome, gallstone and cholecystectomy) known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. History of tuberculosis, any other significant lung diseases like surgeries, asthma, COPD.
4. Upper respiratory tract infections within 14 days of the first study day, or lower respiratory tract infection within 3 months prior to screening.
5. Any clinically significant illness, medical/surgical procedure, or trauma within

4 weeks of the first administration of IMP. 6 Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at screening and first admission to the study unit (first treatment period) as judged by the PI. 7 Any clinically significant abnormal findings in vital signs at screening and first admission to the study unit (first treatment period), as judged by the PI, and defined as:

1. Systolic BP <90 mmHg or ≥140 mmHg and diastolic BP <50 mmHg or

   ≥90 mmHg
2. Heart rate <50 beats per minute [bpm] or >90 bpm Note: Assessments may be repeated once to confirm values. 8 Any clinically significant abnormalities on 12-lead ECG at screening and first admission to the study unit (first treatment period), as judged by the PI, and defined as:

(1) Sick sinus syndrome (2) Arrhythmia (3) Prolonged QT interval corrected using Fridericia's formula (QTcF) > 450 ms (4) Family history of long QT syndrome, persistent or intermittent bundle branch block (BBB), AV block grade II or III 9 Any positive result on screening for serum hepatitis B surface antigen (HBsAg) OR anti-hepatitis B core antigen (HBc) antibody, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody. 10 Has received another new chemical and biologic entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded. 11 Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening. 12 History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to abediterol. 13 Current smokers or those who have smoked or used nicotine products (including e- cigarettes; > 10 pack-year) within the 3 months prior to screening. 14 Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP. 15 Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.

16 Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI or positive screen for drugs of abuse, cotinine, and/or alcohol at screening or on each admission to the Clinical Unit. 17 Subjects with a pregnant partner. 18 Involvement of any AstraZeneca, Parexel or study site employee or their close relatives. 19 Subjects who have previously received abediterol. 20 Judgement by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements. 21 Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Geometric mean ratios and 90% confidence intervals for area under plasma (AUC) for test versus abediterol reference treatments | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To estimate the relative bioavailability of abediterol following inhalation via PARI LC SPRINT nebulizer (2 dose levels) or via OMRON NE-C900-E nebulizer (1 dose level) compared to inhalation via DPI SD2FL (1 dose level)
Geometric mean ratios and 90% confidence intervals for area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC[0-t]) for test versus reference abediterol treatments | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To estimate the relative bioavailability of abediterol following inhalation via PARI LC SPRINT nebulizer (2 dose levels) or via OMRON NE-C900-E nebulizer (1 dose level) compared to inhalation via DPI SD2FL (1 dose level)
Geometric mean ratios and 90% confidence intervals for maximum observed plasma concentration (Cmax) the for test versus reference abediterol treatments | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To estimate the relative bioavailability of abediterol following inhalation via PARI LC SPRINT nebulizer (2 dose levels) or via OMRON NE-C900-E nebulizer (1 dose level) compared to inhalation via DPI SD2FL (1 dose level)

SECONDARY OUTCOMES:
AUC for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
AUC (0-t) for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Cmax for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Area under the plasma concentration-time curve from time zero to 24 hours [AUC (0-24)] for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Maximum concentration (tmax) for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Terminal elimination rate constant (λz) for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Time of last quantifiable plasma concentration (tlast) for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRT) for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) for each abediterol treatment | On Day 1: pre-dose, 5 min [only for DPI], 12, 30, and 45 min, and 1, 2, 4, 6, 8, 12 hours post-dose, on Day 2: 24 and 36 hours post-dose, on Day 3: 48 hours post-dose, on Day 4-7: 72, 96, 120 and 144 hours post-dose.
  To evaluate the PK profile of abediterol when administered via the 3 devices (DPI and 2 nebulisers)
Number of subjects with adverse events | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal electrocardiogram (ECG) | From Screening (Day -28), Day -1 until Day 3
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal telemetry | Day -1, 1 (pre-dose to 12 hours from the start of study drug administration)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal vital signs | From Screening (Day -28) until Day 3
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal physical examination | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal spirometry | At Screening (Day -28) and Day 1
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal taste questionnaire | Day 1
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal White blood cell (WBC) count | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Red blood cell (RBC) count | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Hemoglobin (Hb) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Hematocrit (HCT) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Mean corpuscular volume (MCV) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Mean corpuscular hemoglobin (MCH) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Mean corpuscular hemoglobin concentration (MCHC) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Neutrophils absolute count | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Lymphocytes absolute count | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Monocytes absolute count | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Eosinophils absolute count | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Basophils absolute count | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Reticulocytes absolute count | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal sodium | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal pottasium | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal urea | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal creatinine | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal albumin | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal calcium | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal phosphate | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal glucose (fasting) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal C-reactive protein (CRP) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Alkaline phosphatase (ALP) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Alanine aminotransferase (ALT) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Aspartate aminotransferase (AST) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Total Bilirubin | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Unconjugated bilirubin | Screening (Day -28), Day -1, 1 and 14 days after last dose
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Thyroid-stimulating hormone (TSH) | Screening (Day -28)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal urinalysis (glucose, blood and protein) | Screening (Day -28) and Day -1
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal Gamma glutamyl transpeptidase (GGT) | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects
Number of subjects with abnormal platelet | From Screening (Day -28) until follow-up (14 days after last dose)
  To further assess the safety of single doses administration of abediterol in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med. Rainard Fuhr, Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home